CLINICAL TRIAL: NCT03885622
Title: A Prospective, Multicentre, Cohort Study Assessing the Safety and Efficacy of the ANTHEM™ CR Total Knee System in Patients Following a Total Knee Arthroplasty
Brief Title: Safety and Efficacy of the ANTHEM™ CR Total Knee System
Acronym: Anthem CR
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew Pte Ltd (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: 17-4065-07
Record Dates: First submitted 2019-02-06; First posted 2019-03-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Non-inflammatory Degenerative Joint Disease
Keywords: NIDJD; ANTHEM™ CR Total Knee System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ANTHEM™ CR Total Knee System — The ANTHEM CR Total Knee System is a CE marked device. It is a cruciate retaining (CR) total knee system. It is intended to be used in patients for primary total knee replacement surgery where the posterior cruciate ligament and collateral ligaments remain intact. It is a comprehensive system which allows surgeons to address simple to complex knee arthroplasties.

SUMMARY:
This clinical study will evaluate the short-term (1- and 2-year) and medium term (5-year) safety and performance of the ANTHEM™ CR Total Knee System in patients with non-inflammatory degenerative joint disease of the knee requiring total knee replacement. Clinical, radiographic, Health Economic Outcomes and safety outcomes will be evaluated.

DETAILED DESCRIPTION:
To assess the safety and performance of the ANTHEM™ CR Total Knee System in patients with degeneration of the knee by demonstrating non-inferiority in the revision-free survival rate at 5 years compared to a literature reference rate of 96.6% (Australian Orthopaedic Association annual report 2016).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a candidate for primary total knee arthroplasty due to degenerative joint disease.
2. Subject is willing to sign and date an EC-approved consent form.
3. Subject has posterior cruciate ligament and all collateral ligaments intact in the index joint.
4. Subject is 18 to 75 years old at time of inclusion.
5. Subject plans to be available through ten (10) years postoperative follow-up.
6. Subject agrees to follow the study protocol.
7. Subject has achieved skeletal maturity as deemed by enrolling investigator.

Exclusion Criteria:

1. Subject would receive the ANTHEM™ CR Total Knee System on the affected knee as a revision for a previously failed (TKA) or unicondylar knee arthroplasty (UKA).
2. Subject received TKA on the contralateral knee as a revision for a previously failed TKA or UKA.
3. Subject has a history of patellar fracture, patellectomy, or patello-femoral Instability.
4. Subject has inflammatory arthritis.
5. Subject possesses a contralateral or ipsilateral revision hip arthroplasty.
6. Subject has ipsilateral hip arthritis resulting in flexion contracture.
7. Subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the Investigator:

   * Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty.
   * Contralateral primary TKA or UKA.
8. Inadequate bone stock which would make the procedure unjustifiable including but not limited to: severe osteopenia/osteoporosis or family history of severe osteoporosis/osteopenia as deemed by the enrolling investigator.
9. Subject has collateral ligament insufficiency.
10. Subject has an active infection or sepsis (treated or untreated) or previous intra-articular infections.
11. Subject has presence of malignant tumor, either primary or metastatic, or benign tumor on leg with the knee to be treated.
12. Subject has conditions that may interfere with the TKA survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes mellitus [i.e. not under treatment with oral/injectable medications to control blood glucose levels], fibromyalgia, moderate to severe renal insufficiency or neuromuscular disease).
13. Subject has contralateral lower extremity condition causing abnormal ambulation (e.g. ankle fusion, ankle arthroplasty, previous hip fracture).
14. Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures.
15. Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study, including mental illness, mental retardation, drug or alcohol abuse.
16. Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1.
17. Any subject that meets the definition of a Vulnerable Subject per ISO14155:2011: individual whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 153 subjects undergoing total knee arthroplasty for degenerative joint disease will be implanted with ANTHEM™ CR Total Knee System.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2034-04-03 (Estimated); Study Completion 2034-08-01 (Estimated)

PRIMARY OUTCOMES:
Non-Inferiority 10 years postoperatively | 10 years postoperatively
  Non-inferiority of 10-year implant survivorship of the ANTHEM™ CR Total Knee System in patients undergoing total knee arthroplasty for osteoarthritis compared to reported literature.

SECONDARY OUTCOMES:
Change in implant fixation measured by radiographic assessment | 6 weeks, 1 year, 2 years, and 5 years
  based on comparison of antero posterior and lateral radiographs
Change in bone integrity measured by radiographic assessment | 6 weeks, 1 year, 2 years, and 5 years
  based on comparison of antero-posterior and lateral radiographs
Number of Adverse Events | 6 weeks, 1 year, 2 years, and 5 years
  Number and frequency of all types adverse events
Quality of life measured by EQ-5D-3L | 6 weeks, 1 year, 2 years, and 5 years
  The EQ-5D-3L will be collected at each follow up visit. It consists of two pages - the EQ-5D descriptive system (page one) and the EQ visual analogue scale (EQ VAS) (page two). The descriptive system consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses.
Pain as measured by Knee Society Score (2011 KSS) | 6 weeks, 1 year, 2 years, and 5 years
  This validated tool that combines an objective physician-derived component with a subjective subject-derived component. The objective section rates alignment, instability, joint motion and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ang Sim, M.D., Principal Investigator — Gachon University Gil Medical; Manuj Wadhwa, M.D., Principal Investigator — Ivy Hospital - Ivy Elite Institute of Orthopaedics
Locations (8):
- India (3):
  - Parekhs Hospital, Ahmedabad, Gujarat
  - Aadhar Health Institute, Hisar, Haryana
  - Ivy Hospital - Ivy Elite Institute of Orthopaedics, Mohali, Punjab
- Italy (2):
  - Instituto Clinico Sant'Ambrogio, Milan
  - Istituto Clinico San Siro, Milan
- Westville Hospital, Westville, Durban, South Africa
- South Korea (2):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranam-do
  - Gachon University Gil Medical Center, Incheon, Korea